CLINICAL TRIAL: NCT01416831
Title: Phase II Randomized Study of High Dose Interleukin-2 Versus Stereotactic Body Radiation (SBRT) and High Dose Interleukin-2 (IL-2) in Patients With Metastatic Melanoma
Brief Title: Comparison of High-dose IL-2 and High-dose IL-2 With Radiation Therapy in Patients With Metastatic Melanoma.
Acronym: SBRT/IL-2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Prometheus Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 11-062A
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Results first posted 2022-11-15 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Melanoma
Keywords: metastatic melanoma; IL-2; Interleukin 2; Radiation; Stereotactic Body Radiation Treatment; SBRT; Immunotherapy
MeSH Terms: conditions — Melanoma | interventions — Radiotherapy; Interleukin-2; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: IL-2 Monotherapy (Active Comparator): Patients receive standard high-dose IL-2 therapy, with an opportunity to crossover to the experimental arm if there is disease progression noted after two cycles of high-dose IL-2. Crossover patients will be included in Arm A.
  Interventions: Drug: High-dose IL-2
- Arm B: SBRT + IL-2 (Experimental): Patients will receive two doses of radiation before receiving high-dose IL-2.
  Interventions: Other: Radiation therapy and high-dose IL-2

INTERVENTIONS:
Other: Radiation therapy and high-dose IL-2 — Patients 1 - 20 will receive a single fraction of radiation. Patients 21 through the completion of the study will receive two fractions. The dose for all patients will be 20 Gy per fraction to the prescription line at the edge of the planning treatment volume (PTV) with the last dose delivered on a Friday before IL-2 administration. For patients receiving two radiation doses, the doses can be administered on the Wednesday and Friday before IL-2 starts. Patients who are assigned to IL-2 monotherapy and have progressive disease after two IL-2 cycles are then eligible to receive SBRT before cycle 3 of IL-2 commences, single fraction for patients 1-20 and two fractions for patients 21- end of study.
  Other Names: Interleukin 2; Stereotactic Body Radiation Therapy (SBRT)
  Arms: Arm B: SBRT + IL-2
Drug: High-dose IL-2 — IL-2 will be given on a Monday at a dose of 600,000 IU per kilogram IV every 8 hours for up to 14 doses each cycle. The second cycle is planned 16 days after cycle 1 but may be delayed up to one week to allow toxicity to resolve. The maximum number of doses that can be given during two cycles will be 28 doses. Patients who respond after two cycles can receive 4 more cycles of IL-2. Patients with disease progression after 2 cycles may elect to receive radiation before a 3rd cycle of IL-2. If patients crossover, IL-2 will be given on the Monday following the last dose of radiation, at a dose of 600,000 IU per kilogram IV every 8 hours for a maximum of 14 doses each cycle. Another cycle is planned 16 days after cycle 3 but may be delayed up to one week to allow toxicity to resolve.
  Other Names: Interleukin 2; Stereotactic Body Radiation Therapy (SBRT).
  Arms: Arm A: IL-2 Monotherapy

SUMMARY:
The purpose of this study is compare the response rates in patients with metastatic melanoma treated with high-dose IL-2 to patients treated with high-dose IL-2 along with radiation therapy.

DETAILED DESCRIPTION:
All patients will receive high-dose IL-2. Half the patients enrolled will be randomly selected to receive radiation therapy to up to three tumors prior to receiving high-dose IL-2. Among the first 20 patients enrolled, those assigned to receive radiation will receive a single dose of radiation and for patients 21-44, those assigned to receive radiation will receive 2 doses of radiation.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of melanoma will be required by previous biopsy or cytology.
* Patients must be ≥ 18 years of age.
* Patients must have tumors amenable to SBRT in lungs, mediastinum, chest wall, bones (other than long bones), or liver (inclusive of immediately adjacent masses), 1 - 3 foci; no minimum size, but none greater than 7 cm. Patients may have other metastases but only a maximum of 3 will be treated.
* ECOG performance status of 0-1.
* Women of childbearing potential must have a serum or urine pregnancy test performed within 72 hours prior to the start of protocol treatment. The results of this test must be negative in order for the patient to be eligible. In addition, women of childbearing potential as well as male patients must agree to take appropriate precautions to avoid pregnancy.
* Patients must sign a study-specific consent form.

Exclusion Criteria:

* No metastatic site amenable to SBRT.
* Patients with brain metastases not candidates for radiosurgery.
* Previous radiation to sites proposed for radiation as part of this study.
* Patients with active systemic, pulmonary, or pericardial infection.
* Pregnant or lactating women.
* Evidence of ischemia on exercise tolerance test, stress thallium study, or baseline EKG.
* DLCO, FEV1 or FEV1/FVC less than 70% of predicted due to clinically significant underlying pulmonary disease. For any pulmonary function test values less than predicted values, the PI will review, and document the patient's suitability for high dose IL-2 therapy.
* WBC < 3.0 x 109/L
* Hgb < 9.0 g/dL
* AST/ALT > 3 times the upper limit of the normal range
* total bilirubin > 1.9 g/dL
* creatinine > 1.9 g/dL
* Patient requires chronic steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Curti, M.D., Principal Investigator — Providence Health & Services; Steven K. Seung, M.D., Principal Investigator — Providence Health & Services; Marka Crittenden, MD, PhD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Cancer Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Curti B, Crittenden M, Seung SK, Fountain CB, Payne R, Chang S, Fleser J, Phillips K, Malkasian I, Dobrunick LB, Urba WJ. Randomized phase II study of stereotactic body radiotherapy and interleukin-2 versus interleukin-2 in patients with metastatic melanoma. J Immunother Cancer. 2020 May;8(1):e000773. doi: 10.1136/jitc-2020-000773. PMID 32467299
- [Derived] Sckisel GD, Mirsoian A, Minnar CM, Crittenden M, Curti B, Chen JQ, Blazar BR, Borowsky AD, Monjazeb AM, Murphy WJ. Differential phenotypes of memory CD4 and CD8 T cells in the spleen and peripheral tissues following immunostimulatory therapy. J Immunother Cancer. 2017 Apr 18;5:33. doi: 10.1186/s40425-017-0235-4. eCollection 2017. PMID 28428882

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 63 potential patients were screened for eligibility at Providence Cancer Institute Franz Clinic and Compass Oncology East Clinic from 2011 to 2017.
Pre-assignment Details: Of the 50 patients who signed consent, six were excluded (3 due to rapid melanoma progression during screening, 2 due to cardiac ischemia on exercise tolerance testing, and 1 due to insurance issues). Of the 44 enrolled patients, 20 were assigned to Arm A, and 7 of those patients chose to participate in the optional crossover portion of the study.
Groups:
- Arm B: SBRT + IL-2: Patients 1-20 who are assigned to receive radiation therapy will receive a single dose of radiation before IL-2; patients 21-44 assigned to receive radiation will receive two doses of radiation before receiving high-dose IL-2.
  Radiation therapy and high-dose IL-2: Patients 1 - 20 will receive a single fraction of radiation. Patients 21 through the completion of the study will receive two fractions. The dose for all patients will be 20 Gy per fraction to the prescription line at the edge of the planning treatment volume (PTV) with the last dose delivered on a Friday before IL-2 administration. For patients receiving two radiation doses, the doses can be administered on the Wednesday and Friday before IL-2 starts. Patients who are assigned to IL-2 monotherapy and have progressive disease after two IL-2 cycles are then eligible to receive SBRT before cycle 3 of IL-2 commences, single fraction for patients 1-20 and two fractions for patients 21- end of study.
Period: Cycles 1 & 2 (Weeks 1-14)
Arm/Group | Arm A: IL-2 Monotherapy | Arm B: SBRT + IL-2
Started | 20 | 24
Completed | 19 | 22
Not Completed | 1 | 2
Not completed — Death | 1 | 2
Period: SBRT Crossover Period
Arm/Group | Arm A: IL-2 Monotherapy | Arm B: SBRT + IL-2
Started (Of the 8 patients enrolled into Arm A whose melanoma progressed after the first imaging, 7 agreed to participate in the crossover portion of the study after completion of Cycle 2.) | 7 | 0
Completed | 7 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: IL-2 Monotherapy | Arm B: SBRT + IL-2 | Total
Number analyzed (Participants) | 20 | 24 | 44
Age, Continuous [Mean (Full Range); unit: years] | 57.5 [30 to 82] | 53 [21 to 75] | 57 [21 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 16 | 18 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 24 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 24 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 24 | 44
BRAF Status [Count of Participants; unit: Participants]
  Mutated | 11 | 7 | 18
  Wild Type | 5 | 14 | 19
  Unknown | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Tumor Response of High Dose IL-2 vs. SBRT + High Dose IL-2
Description: Determine the best overall tumor response rate of high dose IL-2 versus SBRT + high-dose IL-2 using RECIST v1.1 assessed by CT/MRI, criteria applied to all target and non-target lesions with the exclusion of sites treated with SBRT. For patients who have SBRT after progression on IL-2 monotherapy, the response rate will be recorded, but not counted as a response for the primary objective.
  Overall response rate (ORR) includes all measurable and non-measurable target lesions except the lesions treated by SBRT, which were assessed separately. Both CT and positron emission tomography imaging were employed to assess response.
  Complete Response: disappearance of all target/non-target lesions and no abnormalities on PET; Partial Response: ≥30% decrease in sum of longest diameter (LD) of target lesions; Progressive Disease: ≥20% increase in sum of LD recorded since tx start or appearance of ≥1 new lesions; Stable Disease: Neither qualifying for PR nor PD since tx started.
Time Frame: At the end of Cycle 2 (Week 14).
Population: There will be a comparison of the overall tumor response of patients receiving one versus two SBRT doses. Responses from patients who participated in the crossover portion of the study were excluded.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: IL-2 Monotherapy | Arm B: SBRT + IL-2
Number analyzed (Participants) | 20 | 24
percentage of participants
  Overall Response Rate (ORR) | 54 | 35
  Complete Response (CR) | 15 | 21
  Partial Response (PR) | 20 | 33
  Stable Disease (SD) | 25 | 21
  Progressive Disease (PD) | 40 | 25

2. Secondary Outcome: Response Rate in Crossover Patients
Description: Measure the response rate of patients who have disease progression after the first IL-2 cycles (using RECIST criteria) who received SBRT prior to cycle 3 of IL-2.
Time Frame: 7 weeks following Cycle 2 (Week 21).
Population: This measure is specifically for patients enrolled into IL-2 monotherapy cohort who then opted for radiation therapy in addition to IL-2.
Measure: Number; unit: Count of participants
Arm/Group | Arm A: IL-2 Monotherapy | Arm B: SBRT + IL-2
Number analyzed (Participants) | 7 | 0
Count of participants
  CR | 1 |
  PR | 2 |
  SD | 0 |
  PD | 4 |

ADVERSE EVENTS:
Time Frame: Screening through Week 7 (or 8 if IL-2 restaging) and during the optional crossover phase, up to 7 weeks.
Description: All adverse events reported during the course of the study.
Groups:
- Arm B: SBRT + IL-2: Patients 1-20 who are assigned to receive radiation therapy will receive a single dose of radiation before IL-2; patients 21-44 assigned to receive radiation will receive two doses of radiation before receiving high-dose IL-2.
  Radiation therapy and high-dose IL-2: Patients 1 - 20 will receive a single fraction of radiation. Patients 21 through the completion of the study will receive two fractions. The dose for all patients will be 20 Gy per fraction to the prescription line at the edge of the planning treatment volume (PTV) with the last dose delivered on a Friday before IL-2 administration. For patients receiving two radiation doses, the doses can be administered on the Wednesday and Friday before IL-2 starts. Patients who are assigned to IL-2 monotherapy and have progressive disease after two IL-2 cycles are then eligible to receive SBRT before cycle 3 of IL-2 commences, single fraction for patients 1-20 and two fractions for patients 21- end of study.
  Patients 25-31 are those who participated in the optional crossover period from Arm A and are included in the at risk figure.
Arm/Group | Arm A: IL-2 Monotherapy | Arm B: SBRT + IL-2
All-Cause Mortality (participants affected / at risk) | 16/20 | 18/31
Serious Adverse Events (participants affected / at risk) | 17/20 | 17/31
Other Adverse Events (participants affected / at risk) | 2/20 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: IL-2 Monotherapy (N=20) | Arm B: SBRT + IL-2 (N=31)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Creatinine Increased (Renal and urinary disorders) | 5 (5) | 9 (11)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (8) | 10 (14)
Hypotension (Vascular disorders) | 13 (19) | 12 (21)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Lymphocyte Count Decreased (Investigations) | 17 (30) | 17 (29)
Platelet Count Decreased (Investigations) | 3 (5) | 4 (4)
Radiation Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (2)
Tachycardia (Cardiac disorders) | 1 (1) | 3 (4)
Acute Ischemic Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Acute Occlusive Thrombus (Vascular disorders) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 3 (3) | 0 (0)
ALT Increased (Investigations) | 2 (2) | 1 (2)
Arthralgias (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bilirubin increased (Investigations) | 6 (7) | 7 (8)
Chest Pain, Severe (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Azotemia (General disorders) | 0 (0) | 1 (1)
Carbon Dioxide Decreased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4) | 5 (8)
Itching (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Left proximal femoral replacement (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (2) | 0 (0)
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Neuropathy, hands (Nervous system disorders) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pulmonary Emboli (Vascular disorders) | 0 (0) | 1 (1)
Rigors (General disorders) | 0 (0) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Systemic Inflammatory Repsonse (Immune system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Troponin Increased (Investigations) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weight Loss (Investigations) | 0 (0) | 1 (1)
White Blood Cells Decreased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: IL-2 Monotherapy (N=20) | Arm B: SBRT + IL-2 (N=31)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alkaline Phosphate Increased (Investigations) | 2 (2) | 0 (0)
ALT (SGPT) Increased (Investigations) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
AST (SGOT) Increased (Investigations) | 2 (2) | 0 (0)
Bilirubin Increased/Elevated (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Capillary leak pulmonary (Vascular disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Creatinine Increased (Investigations) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Drowsiness (Nervous system disorders) | 1 (1) | 0 (0)
Edema, lower extremity (General disorders) | 1 (1) | 0 (0)
Erythroderma (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Mucositis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Myalgias (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Oliguria (Investigations) | 1 (1) | 0 (0)
Pain, abdominal (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pain, knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Dry Desquamation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin, Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vitiligo, upper extremity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vivid Dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Azotemia (General disorders) | 1 (1) | 0 (0)
White Blood Cells Decreased (Investigations) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-05-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT01416831/Prot_SAP_000.pdf
  • Informed Consent Form (2013-05-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT01416831/ICF_001.pdf